CLINICAL TRIAL: NCT03967821
Title: Translation and Validation of the French Quality of Recovery Questionnaire (QoR-15) Postoperative Recovery Assessment Questionnaire
Brief Title: Translation and Validation of the French Quality of Recovery (QoR-15) Questionnaire - Postoperative Recovery Assessment Questionnaire
Acronym: FQoR-15
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC19_0096
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-05

CONDITIONS: Surgery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Each patient complete FQoR-15 questionnaire 3 times (before surgery, on Day 1, on Day 2)

SUMMARY:
Surgery (under general anaesthesia or under loco-regional anaesthesia) is an event that causes stress, anxiety, pain and even minor complications such as nausea or vomiting. Peri-operative management and the psychological support allocated to each patient will have an impact on the hospitalization experience. Many studies have focused on reducing peri-operative mortality (decrease in pain intensity as measured by analog visual scale, decrease in nausea/vomiting frequency, decrease in remobilization time, etc.) but few assessed the overall recovery of patients. there is a desire to improve physical and psychological recovery, with particular attention to the patient's own feelings. It is essential to evaluate our peri-operative management practices based on patient-centred criteria. In this context, the development of a scale for measuring the quality of post-operative recovery appears to be necessary. In 2013, a questionnaire was quickly run (about 2-3 min): the QoR-15 was validated. This questionnaire is reliable, sensitive, easily achievable in clinical practice, not onerous for the patient and provides information on the post-operative recovery perceived by the patient himself.

The QoR-15 was validated in English, then in Danish, Chinese, Portuguese and more recently in Swedish. It has not yet been validated in French and therefore cannot be used in studies on francophone patients.

Investigator goal is to validate a French version of the QoR-15, the FQoR-15.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years old or older)
* Francophones;
* Admitted for any type of scheduled surgery;
* Able to complete the questionnaire upon admission, alone or with the assistance of a third party;
* Agreeing to participate in the study.

Exclusion Criteria:

* Psychiatric or neurological pathology compromising cooperation in the validation protocol of the questionnaire;
* Hospitalized for intracranial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients admitted for any type of scheduled surgery except intracranial
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
To assess the validity of the French version of FQoR-15 to assess post-operative recovery from general or loco-regional anaesthesia | day 2

SECONDARY OUTCOMES:
To ensure the validity of the questionnaire in the context of general anesthesia versus loco-regional anaesthesia | day 2
To assess the validity of the questionnaire specifically in the outpatient sub-population, which will be evaluated by telephone | day 2
to analyze questionnaire validity by type of surgery | day 2

CONTACTS AND LOCATIONS:
Locations (1):
- RINEAU Emmanuel, Angers, France

IPD SHARING:
Plan to Share IPD: No